CLINICAL TRIAL: NCT06424626
Title: A Phase Ib, Open, Mono-center, Dose-reduction Tolerability Study of AK104 or AK112 in Combination With Axitinib in Patients With Metastatic Mucosal Melanoma
Brief Title: A Trial of AK104 or AK112 in Combination With Axitinib in Patients With Metastatic Mucosal Melanoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-043
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2023-12

CONDITIONS: Melanoma; Mucosal Melanoma; Metastatic Melanoma
Keywords: Melanoma; AK104; AK112; Mucosal Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK104 in Combination With Axitinib (Experimental): The planned cohorts in part A were axitinib 5mg twice a day plus AK104 10mg/kg every 3 weeks. A minimum of three patients were initially enrolled at the first dose level. If a dose-limiting toxicity occurred, then the cohort would be expanded to a total of six patients. Responses were evaluated by investigators using both RECIST version 1.1 and Immune-Related RECIST (irRECIST).
  Interventions: Drug: AK104+Axitinib
- AK112 in Combination With Axitinib (Experimental): The planned cohorts in part A were axitinib 5mg twice a day plus AK112 20mg/kg every 3 weeks. A minimum of three patients were initially enrolled at the first dose level. If a dose-limiting toxicity occurred, then the cohort would be expanded to a total of six patients. Responses were evaluated by investigators using both RECIST version 1.1 and Immune-Related RECIST (irRECIST).
  Interventions: Drug: AK112+Axitinib

INTERVENTIONS:
Drug: AK104+Axitinib — Subjects receive AK104 10mg/kg intravenously (IV) every 3-week cycle plus Axitinib until progression.
  Other Names: Cadonilimab
  Arms: AK104 in Combination With Axitinib
Drug: AK112+Axitinib — Subjects receive AK112 20mg/kg intravenously (IV) every 3-week cycle plus Axitinib until progression.
  Other Names: Ivonescimab
  Arms: AK112 in Combination With Axitinib

SUMMARY:
This study was a phase IB, single-center, open-label, two part(part A involved dose reduction, and part B involved cohort expansion) clinical trial evaluating the safety and clinical activity of AK104 or AK112 in combination with axitinib in patients with advanced mucosal melanoma.

DETAILED DESCRIPTION:
The planned cohorts in part A were axitinib 5mg twice a day plus AK104 or AK112 every 3 weeks. A minimum of three patients were initially enrolled at the first dose level. If a dose-limiting toxicity occurred, then the cohort would be expanded to a total of six patients. Responses were evaluated by investigators using both RECIST version 1.1 and Immune-Related RECIST (irRECIST). Patients with progressive disease or an intolerant toxicity were taken off the study. Patients who initially developed progressive disease per RECIST version 1.1 were allowed to continue therapy if the investigator considered patients to be benefiting from the treatment per irRECIST. Any dose-reduction cohort that did not exceed the maximum-tolerated dose could be expanded in part B for additional evaluation of safety and clinical activity. The primary end point of this study was dose-limiting toxicity within the first 4 weeks of treatment with AK104 or AK112 plus axitinib in part A.

ELIGIBILITY:
Inclusion Criteria:

1、18 to 70 years old (at the time consent is obtained). 2、Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures).

3、Have histologically- or cytologically-confirmed diagnosis of Metastatic Mucosal Melanoma.

4、Have a life expectancy of at least 3 months 5、Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 6、Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as determined by the site study team 7、Has adequate organ function as defined by:Absolute neutrophil count ≥ 1,500/µL;Platelets ≥ 100,000/µL;Hemoglobin ≥ 9 g/dL;Crcl ≥ 50ml/min creatinine clearance may be calculated using the institutional/laboratory standard method.Serum total bilirubin ≤ 1.5 x ULN ;Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN ;Albumin ≥28g/L;International Normalized Ratio (INR) and aPTT <1.5 x ULN. Left ventricular ejection fraction ≥50%.

8、Have recovered from the effects of any prior radiotherapy or surgery 9、All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment.

Exclusion Criteria:

1. Prior treatment with anti-PD-1/PD-L1/PD-L2 antibody and Axitinib
2. Is currently participating in a study of an investigational agent or using an investigational device
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy within 2 years prior to the first dose of study treatment
4. Has undergone major surgery within 30 days of Study Day 1
5. Has a known additional malignancy that is progressing or requires systemic treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
6. Has known active central nervous system (CNS) metastases
7. Has carcinomatous meningitis
8. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment NOTE: Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study
9. Has an active infection requiring systemic therapy
10. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected)
11. History of myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or surgery within 12 months prior to day 1 of study treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-21 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 years
  Safety assessments including vital signs, laboratory tests, and adverse event monitoring

SECONDARY OUTCOMES:
Objective Response Rate (ORR) by irRC and RECIST 1.1 | 3 years
  The treatment effect of AK104 or AK112 in combination with axitinib, will be assessed using irRC and RECIST 1.1 to determine tumor response.
Duration of Response (DOR) by irRC and RECIST 1.1 | 3 years
  The treatment effect of AK104 or AK112 in combination with axitinib, will be assessed using irRC and RECIST 1.1 to determine duration of response.
Disease Control Rate (DCR) by irRC and RECIST 1.1 | 3 years
  The treatment effect of AK104 or AK112 in combination with axitinib, will be assessed using irRC and RECIST 1.1 to determine disease control rate.
Time to response (TTR) by irRC and RECIST 1.1 | 3 years
  The treatment effect of AK104 or AK112 in combination with axitinib, will be assessed using irRC and RECIST 1.1 to determine time to response.
Progression-free survival(PFS) by irRC and RECIST 1.1 | 3 years
  The treatment effect of AK104 or AK112 in combination with axitinib, will be assessed using irRC and RECIST 1.1 to determine progression-free survival time.
Overall survival (OS) by irRC and RECIST 1.1 | 3 years
  The treatment effect of AK104 or AK112 in combination with axitinib, will be assessed using irRC and RECIST 1.1 to determine overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No